CLINICAL TRIAL: NCT00153868
Title: Pilot Web-based Study of Functional Status, Symptom Palliation and Quality of Life Benefits Associated With Darbepoetin Alfa (Aranesp®) Administration in Anemic Patients With Cancer.
Brief Title: A Web-based Study of Quality of Life Benefits Associated Aranesp in Anemic Patients With Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Konstantin Dragnev, Associate Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D-0341
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Anemia; Cancer
Keywords: Anemia; Cancer; Quality of life; Web-based; Aranesp; Darbepoetin alfa
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Darbepoetin alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Active Comparator): Darbepoetin alfa 200 mcg with escalation to 300 mcg after 6 weeks (week 7 dose) for non-responders subcutaneously every 2 weeks for 12 weeks (weeks 1, 3, 5, 7, 9, and 11)
  Interventions: Biological: darbepoetin alfa
- 2 (Active Comparator): darbepoetin alfa 300 mcg with escalation to 500 mcg after 6 weeks (week 7 dose) for non-responders subcutaneously every 3 weeks for 12 weeks (weeks 1, 4, 7, and 10)
  Interventions: Biological: darbepoetin alfa

INTERVENTIONS:
Biological: darbepoetin alfa — The allocation to the treatment arms will be dependent on the schedule of chemotherapy (i.e. weekly, every 2 week, or every 4 week chemotherapy schedules will receive a starting dose of 200 mcg darbepoetin alfa and every 3 week chemotherapy schedule will receive a starting dose of 300 mcg). Non-responders are defined as patients who experience <1.0 g/dL increase in hemoglobin concentrations after 6 weeks. Darbepoetin alfa will be held for hemoglobin concentrations >13.0 g/dL.
  Other Names: aranesp

SUMMARY:
This is a web-based pilot study to evaluate the association between the treatment of anemia with darbepoetin alfa (aranesp) and the clinical benefits in symptom palliation, improved functional status and quality of life in patients with cancer. The feasibility of web-based assessments and data capture will be evaluated.

DETAILED DESCRIPTION:
Anemia associated with lung cancer and chemotherapy is an important factor effecting patient symptoms, functional status, and overall quality of life (Groopman and Itri 1999; Langer, Choy et al. 2002). Darbepoetin alfa (Aranesp®) has demonstrated a significant effect upon ameliorating chemotherapy-induced anemia in lung cancer (Vansteenkiste, Pirker et al. 2002; Vansteenkiste, Poulsen et al. 2002). This trial is designed to evaluate the association between the treatment of anemia with darbepoetin alfa and direct electronic capture of clinical benefits in cancer-related symptoms, functional status and overall quality of life. This trial uses a secure web-based design to capture the patient-associated symptoms, functional status and quality of life. This novel secure web-based system was selected to improve the efficiency and quality of clinical data capture. If our hypothesis is correct, treatment with darbepoetin alfa will be associated with improved palliation of cancer-related symptoms, improved functional status, and result in overall benefits to the patient's health-related quality of life. The development of a web-based system to directly capture patient-related symptoms, functional status and quality of life will permit us in the future to conduct a national or international trial addressing the effects of darbepoetin alfa on these factors. If our hypothesis is incorrect, it may be that these parameters are not affected by the correction of anemia with darbepoetin alfa or the measures are not sensitive enough to detect these differences. A notable finding would be a clearly defined improvement in symptom palliation, functional status, and quality of life associated with darbepoetin alfa therapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of non-myeloid cancer (myeloproliferative disorders will be excluded).
* Hemoglobin concentration ≤ 11.0 g/dL.
* Age ≥ 18 years.
* Karnofsky performance status ≥ 60%.
* Anemia predominantly due to cancer or chemotherapy.
* Serum creatinine concentration ≤ 2.0 mg/dL.
* Total serum bilirubin ≤ 1.5 times the upper limit of normal.
* Nutritional status adequate to provide vitamin B12 and folate within the normal limits.
* Capacity to complete the web-based functional status, symptom and quality of life assessments.
* Ability to give informed consent.

Exclusion Criteria:

* Untreated symptomatic primary or metastatic cancer involving the central nervous system.
* History of clinically significant iron deficiency.
* Greater than two red blood cell transfusions within 2 weeks of registration or any red blood cell transfusion within 7 days of registration.
* Received epoetin alfa or darbepoetin alfa therapy within 3 weeks prior to randomization.
* History of a seizure disorder.
* Unstable angina, congestive heart failure (New York Heart Association > class II or known ejection fraction < 40%) or uncontrolled cardiac arrhythmias.
* Uncontrolled hypertension defined as a diastolic blood pressure > 100 mmHg.
* Clinical evidence of active infection or inflammatory diseases such as rheumatoid arthritis. Subjects with active rheumatoid arthritis are excluded.
* Known positive test for human immunodeficiency virus infection.
* Known primary hematological disorder which could cause anemia such as sickle cell anemia.
* Pregnant or breast-feeding.
* Not using adequate contraception if of childbearing potential.
* Known hypersensitivity to any recombinant mammalian-derived product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2003-10; Primary Completion 2007-08-17 (Actual); Study Completion 2007-08-17 (Actual)

PRIMARY OUTCOMES:
A secure web-based assessment of cancer-related symptoms (LCSS), functional status (SF-36), and quality of life (FACT-An and PFS) will be obtained every 2 weeks (weeks 3, 5, 7, 9, 11, and 13). | every 2 weeks (weeks 3, 5, 7, 9, 11, and 13)

SECONDARY OUTCOMES:
A blood sample will be obtained to evaluate hemoglobin concentrations every 2 weeks (weeks 3, 5, 7, 9, 11, and 13). | every 2 weeks (weeks 3, 5, 7, 9, 11, and 13)
A blood sample will be obtained to evaluate plasma cytokines every 4 weeks (weeks 5, 9, and 13). | every 4 weeks (weeks 5, 9, and 13)

CONTACTS AND LOCATIONS:
Overall Officials: James R Rigas, MD, Principal Investigator — Norris Cotton Cancer Center
Locations (1):
- Norris Cotton Cancer Center, Lebanon, New Hampshire, United States